CLINICAL TRIAL: NCT06273813
Title: A Phase 1 Safety, Tolerability and Pharmacokinetic Study of NOV-1776 Compared to Ketorolac Tromethamine IV in Adult Healthy Volunteers and Gout Patients
Brief Title: Treatment of Topical Ketorolac Gel in Acute Gouty Flare
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novilla Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NOV-1776-CL-101
Record Dates: First submitted 2024-02-15; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Acute Gouty Arthritis; Acute Pain; Gout Flare
Keywords: ketorolac; topical; intravenous
MeSH Terms: conditions — Acute Pain | interventions — Ketorolac Tromethamine

STUDY DESIGN:
Intervention Model Description: All cohost 1 subjects receive single ketorolac tromethamine injection, followed by escalating doses of ketorolac tromethamine gel Cohort 2 and 3 subjects receive doses of ketorolac tromethamine gel for 5 days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ketorolac tromethamine (Experimental): Cohort 1 - All subjects receive one Ketorolac tromethamine injection, followed by Ketorolac tromethamine gel topical Cohort 2 and 3 - Ketorolac tromethamine gel topical
  Interventions: Drug: Ketorolac Tromethamine 15 MG/ML; Drug: Ketorolac Tromethamine

INTERVENTIONS:
Drug: Ketorolac Tromethamine 15 MG/ML — Single intravenous administration of Ketorolac Tromethamine injection in Cohort 1 on day 1
Drug: Ketorolac Tromethamine — Three doses of topical ketorolac tromethamine over the course of 1 day, 6 hours apart for each of 3 subsequent treatment periods in cohort 1 Three doses of Ketorolac Tromethamine, 6 hours apart, over the course of 5 days in cohorts 2 and 3

SUMMARY:
This study will be a phase 1, open-label, bioavailability, safety and PK study of topically applied transcutaneous ketorolac tromethamine gel 12.5% (/w) (NOV-1776) versus intravenous administration of approved ketorolac tromethamine injection, USP (15mg/mL) comparator in healthy volunteers, including an evaluation of safety, tolerability, and efficacy in gout participants with flare-up.

DETAILED DESCRIPTION:
Participants will be in the age range of 18 - 64 years of age (Cohort 1) and 18 - 70 years of age (Cohorts 2 and 3). This study will be conducted in three consecutive cohorts (see Figure 1). Cohorts 1 and 2 is conducted inpatient, while Cohort 3 is conducted outpatient.

- Cohort 1: Open-label, single-day, multiple-dose (three doses), in approximately 8 adult healthy volunteers. Study participants will be admitted to the clinic and receive one intravenous dose of ketorolac tromethamine injection, USP over the course of one day for one treatment period, and three doses of topical drug product over the course of 1 day, 6 hours apart for each of 3 subsequent treatment periods of this Cohort 1. The next dose begins after a 2-day wash-out period, and there are three dose levels for the topically applied transcutaneous ketorolac tromethamine gel 12.5% (w/w) (NOV-1776) to be compared to one intravenous administration of 2 ml of ketorolac tromethamine injection, USP (5 mg/mL).

Safety Review Committee meeting to review Cohort 1 data and approve continuance to Cohort 2.

* Cohort 2: Open-label, 1-arm, 5-day, multiple-dose PK, safety in approximately 12 adult healthy volunteers at the maximum tolerated dose demonstrated by Cohort 1. Study participants will be admitted to the clinic and receive three doses of drug product, 6 hours apart, over the course of 5 days. Cohort 1 participants are eligible to participate in Cohort 2. Safety Review Committee meeting to review Cohort 1 and 2 data and approve continuance to Cohort 3.
* Cohort 3 will be an open-label, 1-arm, 5-day, multiple-dose safety, toleration, and efficacy design in 10 adult gout participants with flare-up

ELIGIBILITY:
Inclusion Criteria:

Cohorts 1 and 2

* Evidence of a personally signed and dated informed consent form (ICF) in English
* Healthy study participants who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures,
* Body mass index (BMI) from 18.0 to 32.0 kg/m2, inclusive; and body weight of at least 50 kg (110 lbs) and Resting supine systolic blood pressure from 90 to 140 mmHg and supine diastolic blood pressure from 40 to 90 mmHg
* Male participants must agree to utilize a barrier contraceptive method for the duration of the study and agree to avoid sperm donation for at least 90 days after completing study participation and female participants must be of non-childbearing potential (defined as either surgically sterile or at least 1 year post-menopausal; post- menopausal is defined as no menses for 12 months and confirmed by FSH level ≥ 40 mIU/mL); or must be using a highly effective method of contraception

Cohort 3 - additional requirements

- Medical diagnosis of gout for at least 2 years and1 - 2 acute gout flare-ups within the last 12 months

Exclusion Criteria:

Cohorts 1. 2 and 3

* Presence or history of any disorder that may prevent the successful completion of Cohort 1 [or Cohort 2, as appropriate]
* Allergy or sensitivity to non-steroidal anti-inflammatory drugs (NSAIDs), ketorolac tromethamine, or any components of the formulation and /or history of significant allergies and hypersensitivity reactions (hives, breathing difficulty, etc.) to aspirin or any other medications, either prescription or nonprescription, including dietary supplements or herbal medications.
* A clinically significant history of or current abnormality or disease of any organ system, including renal, hepatic, gastrointestinal (e.g., bleeding, ulcers, perforation), cardiovascular (e.g., cardiovascular thrombotic events, myocardial infarction, stroke) pulmonary (including chronic asthma), endocrine (e.g., diabetes), central nervous system, hematologic system (e.g., bleeding disorders), psychiatric disease, seizure, epilepsy, severe head injury, multiple sclerosis, or other known neurological conditions, or recent surgery that the Investigator deems clinically significant.
* History or recent occurrence of clinically significant skin disorders (including photosensitivity reactions, eczema, and psoriasis) or any surgical or medical condition or skin modification at the site of drug application that may interfere with the absorption, distribution, metabolism or excretion of the test article.
* Hemoglobin < 13.2 g/dL or < 132 g/L (males) and < 11.7 g/dL or < 117 g/L (females); Hematocrit < 38.5% (males) and < 35% (females) platelet count < 100,000 platelets per microliter (males and females); at Screening
* Uncontrolled hypertension with consistent blood pressure higher than 140 / 90 mmHg.
* within 7 days prior to study enrollment, acute illness (e.g., nausea, vomiting, fever, or diarrhea), use of any prescription OTC or dietary or herbal supplements, including ketorolac tromethamine
* within 60 days prior to study enrollment, plasma or blood donation
* within 90 days prior to study enrollment, use of hepatic or renal clearance altering agents (e.g., erythromycin, cimetidine, barbiturates, phenothiazines, St. John's Wort, etc.)
* Positive finding on urine drug screen ( (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, cotinine, methadone, and opiates or other substances deemed inappropriate); Positive serological findings for any of the following: Human Immunodeficiency Virus (HIV), Hepatitis B surface antigen, Hepatitis C antibody, or Hepatitis A IgM tests at Screening.
* Female participants who are pregnant or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | 15 days
  Assessment of adverse events
Area Under the Plasma Concentration Versus Time Curve (AUC) of topical ketorolac tromethamine | 15 days
  Assessment of bioavailability of topical ketorolac tromethamine

CONTACTS AND LOCATIONS:
Overall Officials: Novotech CRO, Study Director — Novotech
Locations (2):
- Australia (2):
  - Paratus Clinical,, Blacktown
  - Linear Clinical Research Ltd, Nedlands

IPD SHARING:
Plan to Share IPD: Undecided